CLINICAL TRIAL: NCT05947708
Title: A Post-Market, Single Blind, Randomized Clinical Prospective Study on Intradialytic Symptoms in Subjects Treated With Qd 500vs Qd 300
Brief Title: The Study of Intradialytic Symptoms in Subjects Treated With Qd 500vs Qd 300
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Outset Medical (Industry)
Collaborators: White Plains Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-03
Record Dates: First submitted 2023-06-21; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-06

CONDITIONS: End Stage Renal Disease on Dialysis
Keywords: Hemodialysis; Flow Rate

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to either arm at a 1:1 ratio using excel's RANDBETWEEN function. Subjects will be randomly assigned a 0 or a 1. Subjects that are assigned '0' will go to Group 1, and subjects that are assigned '1' will go to Group 2.
Who Masked: Participant
Masking Description: Only Subjects will be blinded to the dialysis device Qd.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- High FLow Rate (Active Comparator): Flow Rate of 500ml/min or higher
  Interventions: Device: Dialysate Flow Rate
- Low Flow Rate (Active Comparator): Flow Rate of 300ml/min
  Interventions: Device: Dialysate Flow Rate

INTERVENTIONS:
Device: Dialysate Flow Rate — Hemodialysis is completed with dialysate being used at differing flow rates. Flow rates will be modified to see if this is a causal factor in post-dialysis recovery.

SUMMARY:
Study Goal is to determine the impact of dialysate flow rate (Qd) on Subject reported dialysis related symptoms and on time to recovery post dialysis.

DETAILED DESCRIPTION:
The objective of this study is to determine if Subjects who report dialysis symptoms while meeting adequacy (as determined by Kt/V of 1.2 or greater) on thrice weekly dialysis or who have a recovery time of at least 4 hours when treated on a conventional, i.e. non Tablo, hemodialysis device feel better with a reduced dialysate flow rate of 300ml/min based on an assessment of time to recovery post dialysis and Subject reported symptoms via a modified weekly ESAS survey.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided informed consent and has signed a Health Insurance Portability and Accountability Act of 1996 (HIPAA) compliant authorization statement.
2. Subject is at least 18 of age.
3. Subject has end stage renal disease (ESRD) adequately treated with thrice weekly dialysis.
4. Subject is currently stable on dialysis for at least 3 months on a conventional dialysis machine and Qd of 500ml/min or higher with no change in the following dialysis prescription parameters over that time: Qb, Qd, Dialyzer, Time.
5. Subject has a baseline Kt/V of greater than 1.2.
6. Subject has a stable vascular access.
7. Subject reports time to recovery of more than 4 hours or a modified ESAS with at least 5 symptoms of which at least 2 are rated as moderate (rating of 4-6) or severe (rating of 7-10).

Exclusion Criteria:

- 1. Subject is unable to complete the questionnaires. 2. Subject is pregnant or planning to become pregnant. 3. Subject is scheduled for a change in modality or expected kidney transplant in the next 3 months.

4. Any other documented condition that the Investigator feels would prevent the Subject from successful inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Adequacy of Chronic Dialysis | 4 weeks
  Adequacy (as determined by Kt/V of 1.2 or greater) of patients treated with chronic (3x/wk), dialysis or who have a recovery time of more than 4 hours, when treated on a Tablo hemodialysis device versus conventional, i.e. non Tablo, hemodialysis device.
Post-Treatment Symptomology | 0-24 Hours
  Occurrence Rate of post-treatment symptoms (24hrs) when treated with a reduced dialysate flow rate of 300ml/min, based on an assessment of time to recovery post dialysis when using Tablo hemodialysis device, when compared to occurrence of post-treatment symptoms (24hrs) reported with dialysate flow rates ≥ 500 ml/min on conventional dialysis machines.

SECONDARY OUTCOMES:
Weekly Modified Edmonton Symptom Assessment System (ESAS) | 4 weeks
  Patient's assessment of symptom severity (i.e.,pain, tiredness, drowsiness, nausea, shortness of breath, appetite, depression, anxiety, and wellbeing).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Gunter, Study Director — Outset Medical
Locations (1):
- Outset Medical, San Jose, California, United States

IPD SHARING:
Plan to Share IPD: No
The data derived from this clinical study will be shared via peer-reviewed journals and/or abstracts to nephrology centered conferences.

DOCUMENTS (1):
  • Study Protocol (2019-09-15): https://cdn.clinicaltrials.gov/large-docs/08/NCT05947708/Prot_000.pdf